CLINICAL TRIAL: NCT00071630
Title: Process as a Predictor of Outcomes in CBT for Youth
Brief Title: Therapeutic Processes and Treatment Outcome in Adolescents With Anxiety Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH064484 (NIH); R01MH064484 (NIH); DSIR CT-S
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2008-09

CONDITIONS: Anxiety Disorders
Keywords: Adolescent
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to examine the relationship between different aspects of cognitive behavior therapy (CBT) and treatment outcome.

DETAILED DESCRIPTION:
Anxiety disorders are common among children; if untreated, they can negatively affect children's lives. Evidence suggests that CBT can benefit children with anxiety disorders, but the causal mechanisms between therapy and beneficial outcomes have not been thoroughly investigated.

Audio and videotaped sessions of children currently receiving CBT and those who received CBT in previous trials will be examined. Various rating scales will be used to rate therapeutic alliance, child involvement, and therapist flexibility for each session of CBT. To evaluate potential process variables that contribute to participant drop-out, this study will compare the early process variables for children who complete treatment and for those who discontinue treatment.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of separation anxiety disorder, generalized anxiety disorder, or social phobia
* At least one English-speaking parent

Exclusion criteria:

* IQ < 80
* Psychotic symptoms

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130
Dates: Start 2002-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (2):
- Temple University, Philadelphia, Pennsylvania, United States
- Macquarie University, Sydney, New South Wales, Australia